CLINICAL TRIAL: NCT00068497
Title: Single Agent ZD-1839 (NSC-715055, IND-61187) in Patients With Advanced Head and Neck Carcinoma or Non-Small Cell Lung Cancer Aged 75 Years and Older (and in a Cohort of Patients 50 Years Old and Younger)
Brief Title: Gefitinib in Treating Patients With Metastatic or Unresectable Head and Neck Cancer or Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03171; S0322; U10CA032102 (NIH); CDR0000322890 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Anaplastic Thyroid Cancer; Insular Thyroid Cancer; Metastatic Parathyroid Cancer; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Non-small Cell Lung Cancer; Recurrent Parathyroid Cancer; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Thyroid Cancer; Recurrent Verrucous Carcinoma of the Larynx; Stage III Follicular Thyroid Cancer; Stage III Papillary Thyroid Cancer; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Larynx; Stage IIIB Non-small Cell Lung Cancer; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Non-small Cell Lung Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Adenoid Cystic Carcinoma of the Oral Cavity; Stage IVA Basal Cell Carcinoma of the Lip; Stage IVA Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Follicular Thyroid Cancer; Stage IVA Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IVA Lymphoepithelioma of the Oropharynx; Stage IVA Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IVA Mucoepidermoid Carcinoma of the Oral Cavity; Stage IVA Papillary Thyroid Cancer; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Adenoid Cystic Carcinoma of the Oral Cavity; Stage IVB Basal Cell Carcinoma of the Lip; Stage IVB Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Follicular Thyroid Cancer; Stage IVB Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IVB Lymphoepithelioma of the Oropharynx; Stage IVB Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IVB Mucoepidermoid Carcinoma of the Oral Cavity; Stage IVB Papillary Thyroid Cancer; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Adenoid Cystic Carcinoma of the Oral Cavity; Stage IVC Basal Cell Carcinoma of the Lip; Stage IVC Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Follicular Thyroid Cancer; Stage IVC Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IVC Lymphoepithelioma of the Oropharynx; Stage IVC Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IVC Mucoepidermoid Carcinoma of the Oral Cavity; Stage IVC Papillary Thyroid Cancer; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Thryoid Gland Nonmedullary Carcinoma; Thyroid Gland Medullary Carcinoma; Tongue Cancer; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Parathyroid Neoplasms; Esthesioneuroblastoma, Olfactory; Carcinoma, Non-Small-Cell Lung; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Carcinoma, Medullary; Tongue Neoplasms | interventions — Gefitinib

ARMS (1):
- Treatment (gefitinib) (Experimental): Patients receive oral gefitinib on day 1 and then daily beginning on day 8. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: gefitinib — Given orally
  Other Names: Iressa; ZD 1839

SUMMARY:
This phase I trial is studying the side effects of gefitinib in treating patients with metastatic or unresectable head and neck cancer or non-small cell lung cancer. Gefitinib may stop the growth of cancer cells by blocking the enzymes necessary for their growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of enrolling patients ages 75 years or older and 50 years and younger with metastatic or unresectable head and neck cancer or non-small cell lung cancer, to a structured pilot study that includes pharmacokinetic sampling in a special patient population.

II. To preliminarily compare the ZD-1839 peak concentration level, elimination half-life and steady state level between the two patient age groups.

OUTLINE: This is a pilot, multicenter study. Patients are stratified according to age (75 years and over vs 50 years and under)

Patients receive oral gefitinib on day 1 and then daily beginning on day 8. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed for 30 days and then for up to 3 years after study registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed head and neck carcinoma or non-small cell lung cancer which is metastatic or unresectable for which standard curative or palliative measures do not exist or are no longer effective or are likely to be as effective as ZD1839; patients with known brain metastases are only eligible if their brain metastases have been treated and if in the opinion of the treating physician they are stable
* Patients must be 75 years or older, or 50 years of age or younger
* Serum creatinine =< the institutional upper limit of normal
* Bilirubin =< the institutional upper limit of normal
* SGOT or SGPT =< 2.5 x the institutional upper limit of normal; SGOT and SGPT could be =< 5 x the upper limit of normal if the patient has liver metastases as long as the bilirubin is normal
* AGC of >= 1,500/ul
* Platelet count of >= 100,000/ul
* Patients requiring agents that induce CYP3A4 are excluded from the study, at the present time, agents known to induce CYP3A4 include the antibiotics nafcillin and rifampin, the anticonvulsants carbamazepine, phenobarbital, phenytoin, oxcarbazepine, fosphenytoin and primidone as well as St. John's Wort, rifabutin, rifapentine and modafinil
* Patients may or may not have received prior chemotherapy; patients must not have a curative option and in the opinion of the treating physician there is no other treatment option likely to provide greater benefit; patients must not have received prior treatment with EGFR inhibitors; patients must have recovered from the effects of prior therapy; all prior therapies must be documented
* Patients must have a performance status of 0-2 by Zubrod standards
* Patients must not be planning to receive concurrent radiation therapy, hormone therapy, chemotherapy or immune therapy for malignancy while receiving protocol treatment
* Patients must agree to undergo pharmacokinetic sampling and sample submission
* Patients known to be HIV positive and receiving retroviral therapies are not eligible
* Patients with any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac or infection) are not eligible
* Patients must be able to swallow oral medication in pill form; patients may not receive study medication through a feeding tube
* A baseline slit lamp examination is NOT required; however, patients with eye symptoms (eye pain, tearing, redness, vision problems) or known eye disorders should be evaluated by an ophthalmologist/optometrist prior to registration and the results documented on the toxicity form in the notes section
* Patients must not be pregnant or nursing; patients of reproductive potential must have agreed to use an effective contraceptive method
* If day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day
* In calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday four weeks later would be considered day 28; this allows for efficient patient scheduling without exceeding guidelines
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-08; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrolling patients aged 75 or older and 50 or younger to the study setting | 1 year
Peak ZD1839 concentration level | Up to 3 years
Elimination half-life | Up to 3 years
Toxicity rates between the two age groups by CTCAE version 3.0 | Up to 3 years
Responses observed | Up to 3 years
  Will be reported separately for the two tumor types, i.e., head and neck vs. lung cancer, with 95% confidence intervals for the estimated response rates.
Survival for each tumor type | Up to 3 years
  Kaplan-Meier curves will summarize with median estimates and associated 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Shirish Gadgeel, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States